CLINICAL TRIAL: NCT00143572
Title: Phase I Study of Combination Treatment With Hydroxyurea and Magnesium Pidolate in Patients With Sickle Cell Disease
Brief Title: Use of Hydroxyurea and Magnesium Pidolate for Treatment of Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUMG1
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2010-02

CONDITIONS: Anemia, Sickle Cell
Keywords: Hematologic Diseases; Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases | interventions — Pyrrolidonecarboxylic Acid; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Magnesium Pidolate, Hydroxyurea

INTERVENTIONS:
Drug: Magnesium Pidolate, Hydroxyurea — Intervention Description: Mg pidolate in combination with HU in patients with sickle cell disease who have been on a therapeutic dose (15-30 mg/kg/day) of HU for at least 6 months. Mg pidolate will be given at an initial dose of 0.6 mEq/kg/day divided into 2 daily doses for the first cohort of patients. This dose will be escalated for the subsequent patient cohorts as defined by a classic Phase I design (according to toxicity).

SUMMARY:
The purpose of this study is to estimate the MTD of Mg pidolate in combination with HU in patients with sickle cell disease who have been on a therapeutic dose (15-30 mg/kg/day) of HU for at least 6 months.

DETAILED DESCRIPTION:
This is a Phase I clinical trial evaluating the combination of hydroxyurea and magnesium pidolate for patients with sickle cell disease with either hemoglobin SS disease or hemoglobin S beta thalassemia. Hydroxyurea and magnesium pidolate will be tested in pediatric and adolescent patients with sickle cell disease who already have been treated with hydroxyurea for a minimum of six months. Magnesium pidolate will be given in combination with hydroxyurea for six months. In successive small groups of patients, the dose of magnesium will be increased in order to eventually determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) for magnesium when given in combination with hydroxyurea. The maximum tolerated dose is the highest drug dose that can be given safely to participants. The dose limiting toxicity is determined when drug side effects prevent an increase in dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 3 years and < 15 years at the time of study enrollment
2. Diagnosis of Hb SS or Hb S beta thalassemia
3. Hydroxyurea treatment for at least 6 months prior to study entry at dose of 15 - 30 mg/kg/day
4. Compliance with taking HU treatment of at least 70 % for 6 months prior to study entry

Exclusion Criteria:

1. Red blood cell transfusion within the last 3 months resulting in a level of Hb A of 10% or more
2. Pregnancy or unwillingness to use effective birth control in sexually active subjects (females who state that they are sexually active)
3. Renal dysfunction defined by a serum creatinine greater than 1.5 times the upper limit of normal for age
4. Liver dysfunction defined by an ALT greater than twice the upper limit of normal for age
5. Concomitant usage of an "antisickling" agent other than hydroxyurea
6. Current use of Mg containing drugs
7. Iron deficiency, defined by serum ferritin ≤ 10 ng/ml
8. Concomitant chronic illness other than sickle cell anemia

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2004-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose of magnesium pidolate in combination with hydroxyurea in patients with sickle cell disease who have been on a therapeutic dose of hydroxyurea for at least six months. | Every 2 weeks for first 8 weeks; then every 4 weeks

SECONDARY OUTCOMES:
To document the toxicity of the combination of hydroxyurea and magnesium pidolate. | Every 2 weeks for first 8 weeks; then every 4 weeks
To investigate the effect of the combination of hydroxyurea and magnesium on hematological parameters and red cell metabolism. | 3 months, 6 months, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Winfred Wang, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org